CLINICAL TRIAL: NCT07178522
Title: A Prospective, Open-label, Multi-center, Phase 3 Study to Evaluate the Immunogenicity and Safety of an Inactivated EV71 Enterovirus Vaccine (Envacgen®) in Children Aged 6 to <10 Years Compared to Children Aged 2 to <6 Years
Brief Title: A Study to Evaluate the Immunogenicity and Safety of an EV71 Vaccine (Envacgen®) in Children Aged 6 to <10 Years Compared to Children Aged 2 to <6 Years
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CT-EV-32
Record Dates: First submitted 2025-08-21; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Enterovirus 71 Inactivated Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children Aged 6 to <10 Years (Experimental): EV71 Vaccine (Envacgen®)
  Interventions: Biological: Envacgen®
- Children Aged 2 to <6 Years (Active Comparator): EV71 Vaccine (Envacgen®)
  Interventions: Biological: Envacgen®

INTERVENTIONS:
Biological: Envacgen® — Subjects are to receive a 0.5 mL IM injection of Envacgen®. Study drug is administered on Day 1 and Day 57 of the study.

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of EV71 vaccine (Envacgen®) in Children Aged 6 to <10 Years compared to Children Aged 2 to <6 Years.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center, phase 3 study. Participants will receive the first IM injection of study vaccine on Day 1 and will receive a second dose 56 days later. The last study visit is on Day 237 when participants will be contacted via telephone to assess for adverse events .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged 2 to <10 years as established by medical history and clinical examination.
2. Subject and/or the subject's parent/guardian is able to understand and sign the ICF.

Exclusion Criteria:

1. Has poor venous access.
2. Currently has a fever defined as ear/rectal temperature ≥ 38°C or axillary temperature ≥ 37.5 °C within 2 days before the time of planned vaccination.
3. Has had previously known exposure to EV71 or has received EV71 vaccine.
4. Has a history of herpangina or HFMD associated with enterovirus infection in the past 28 days before the date of planned study drug vaccination.
5. Has been diagnosed with a significant neurological, pulmonary, cardiovascular, hematological, hepatic, or renal disorder.
6. Has a history of hypersensitivity to vaccines, or a history of allergic disease or reactions likely to be exacerbated by any component or any residual trace components such as formaldehyde of the Envacgen® vaccine.
7. Has used any investigational/nonregistered product (including drug, vaccine, or invasive medical device) within 28 days before study vaccination or plans to use any of them during the study period.
8. Has confirmed or suspected autoimmune disorder or immunodeficiency.
9. Has been administered or plans to be administered with any licensed live attenuated vaccine within 14 days before or after each study vaccination.
10. Has used immunoglobulins via intravenous route or any blood products within 11 months before vaccination or plans to use any of them during the study period.
11. Has received immunosuppressant, cytotoxic drug, corticosteroid (including prednisolone ≥ 0.5 mg/kg/day or equivalent), immunomodulator or acetylsalicylic acid for > 14 days within 6 months before the first vaccination or plans to use any of them during the study period. (Inhaled and topical steroids are allowed).
12. Has any medical or psychiatric condition that is a contraindication to protocol participation based on the judgment of the Investigator.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 378 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of Envacgen® | Day 1 to 28 days after the second vaccination.
  1. Geometric Mean Titer (GMT) of Neutralizing Antibody (NTAb) Measurement of NTAb titers against EV71 at 28 days after the second dose of Envacgen® in children aged 6 to <10 years (Old group) compared with children aged 2 to <6 years (Young group).
  2. Seroresponse Rate (SRR) of Neutralizing Antibody (NTAb) Percentage of participants with seroresponse (defined as at least a four-fold increase from baseline in NTAb titers) at 28 days after the second dose of Envacgen® in children aged 6 to <10 years (Old group) compared with children aged 2 to <6 years (Young group).
Incidence of Adverse Events(AEs) [Safety] | Day 1 to 28 days after the second vaccination.
  Number and percentage of participants in the Old group (6 to <10 years) and Young group (2 to <6 years) with any reported adverse events within 28 days after vaccination with Envacgen®.

SECONDARY OUTCOMES:
Incidence of Adverse Events(AEs) [Safety] | Day 1 to 180 days after the second vaccination.
  Number of participants with any adverse events (AEs) reported during the study period.

OTHER OUTCOMES:
Immunogenicity of Envacgen® for cross-reaction | Day 1 to 28 days after the second vaccination.
  GMT of neutralizing antibodies against heterologous EV71 genotypes at 28 days after the second dose of Envacgen® in children aged 6 to <10 years (Old group) and children aged 2 to <6 years (Young group).

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Hospital Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No